CLINICAL TRIAL: NCT03618927
Title: A Program Evaluation of an In-school Daily Physical Activity Initiative for Children and Youth
Brief Title: Program Evaluation of an In-school Daily Physical Activity Initiative
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Start2Finish (Unknown); Hamilton-Wentworth Catholic District School Board (Unknown)
Responsible Party: Principal Investigator, John Cairney, Professor, University of Toronto
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INCH_S2F
Record Dates: First submitted 2018-07-24; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Physical Activity; Children, Only
Keywords: intervention; health policy; psychosocial health; education
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily physical activity intervention (Experimental): The intervention consisted of a DPA program designed by a national organization with expertise in school-based physical activity programming and delivered in school by teachers. The program was offered to students in grades 4 through 8 and consisted of 20 minutes of structured DPA in school for 20 consecutive weeks. The DPA activities included jumping jacks, squats, running and other body weight exercises.
  Interventions: Behavioral: Daily physical activity intervention
- Control - treatment as usual (No Intervention): Participants in control classes completed regular school activities as per the Ontario curriculum.

INTERVENTIONS:
Behavioral: Daily physical activity intervention
  Arms: Daily physical activity intervention

SUMMARY:
The school system is one setting in which children's physical activity levels may be increased through daily physical activity (DPA) policies and initiatives. Adherence to DPA policies is typically poor and results are limited in regard to the associated benefits for participating children. Therefore, the purpose of this study was to evaluate a range of psychosocial outcomes following a community-led, in-school DPA initiative for 9-14 year old children and youth. This program evaluation examined the impact of a DPA program consisting of 20 minutes of teacher-led DPA for 20 consecutive weeks. Student outcomes were measured using a questionnaire administered at three time points: baseline, mid-intervention, and post-intervention. A teacher questionnaire regarding program adherence and student behaviour was completed at post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participants will include males and females between the ages of 9-14.
* Participants must be enrolled in one of 30 elementary school classes across the participating seven elementary schools.
* Participants need to be able to read and write in English

Exclusion Criteria:

* Participants not enrolled in one of the participating classes.
* Unable to read and write in English.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 362 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Change in self-esteem from baseline to 20-weeks | Change from baseline to 20-weeks
  Measured using the Rosenberg Self-Esteem Scale. This is a 10-item measure that has shown to have good construct validity in children. The scale is scored on a four-point Likert-type scale ranging from 0 (Strongly Disagree) to 3 (Strongly Agree). An example item is "On the whole, I am satisfied with myself." Items 2, 5, 6, 8, 9 are reverse scored. The scores for the 10 items are then summed, with higher scores indicating higher self-esteem.
Change in grit from baseline to 20-weeks | Change from baseline to 20-weeks
  Assessed with the 8-item Short Grit Scale for Children. The items are scored on a five-point Likert-type scale ranging from 1 (Not at all like me) to 5 (Very much like me). An example item is "New ideas and projects sometimes distract me from previous ones." Items 1,3,5,6 were reversed scored and all items were summed with higher scores indicating better results.
Change in Global Happiness from baseline to 20-weeks | Change from baseline to 20-weeks
  Measured using the 4-item Subjective Happiness Scale. The scale is scored on a seven-point Likert-type scale. Each item has its own stem and anchors ranging from 1 to 7. An example item stem is "In general I consider myself…" with 1 anchored as Not a very happy person and 7 anchored as A very happy person. The scale has demonstrated good psychometric properties in children and adolescents. The sum of scores is divided by four with a higher score indicating a greater level of happiness.
Change in Commitment to School from baseline to 20-weeks | Change from baseline to 20-weeks
  Assessed with 5 items drawn from the 10-item Commitment to School scale. The scale consists of 10-items scored on a four-point Likert-type scale ranging from 1 (Strongly Disagree) to 4 (Strongly Agree). A subset of five-items was selected, scored on a five-point Likert-type ranging from 1 (Not at all true for me) to 5 (Really true for me). An example item is "You try really hard at school." The 5 items were summed with higher score indicating greater commitment to school.
Change in Sense of Belonging at School from baseline to 20-weeks | Change from baseline to 20-weeks
  Measured using the 5-item short form version of the Sense of Belonging Scale. An example item is "I feel comfortable at my school." Two items were reverse scored, and the items were summed with higher scores indicating a greater sense of belonging at school.
Change in Physical Activity from baseline to 20-weeks | Change from baseline to 20-weeks
  Assessed with the Physical Activity Questionnaire for Older Children (PAQ-C). The PAQ-C was designed for children in grades 4-8 who have recess as a regular part of their school week. The PAQ-C is a 9-item 7-day recall instrument that has been shown to have good psychometric properties. We omitted the first item from this questionnaire because it asked about the types of physical activity performed, and we were interested only in overall levels of participation. An example item is "In the last 7 days, what did you do most of the time at recess?" The items were averaged together to generate a total score, with higher scores indicating higher levels of participation in physical activity.
Change in Self-efficacy from baseline to 20-weeks | Change from baseline to 20-weeks
  Self-efficacy for engaging in physical activity, sports, and active play was assessed using a three-item scale adhering to recommendations by Bandura for assessing self-efficacy. Each item was prefaced with the stem "I am confident in my ability to engage in…" The individual items were "Physical activity (e.g., running, yoga, skating)," "Sports (e.g., soccer, baseball, ultimate Frisbee)," and "Activity play (e.g., playing with friends at recess or after school)." Following guidelines provided by Bandura, participants rated their confidence for each item using an 11-point scale (0=not confident, 10=totally confident). A generalized task self-efficacy overall score was computed by averaging the ratings for each item to produce a scale value out of 10. Higher scores indicate more favorable self-efficacy.

SECONDARY OUTCOMES:
Intervention adherence | 20-weeks
  Assessed by teacher questionnaire: "On average, how many days per week did your students participate in the program?". A higher score indicates greater adherence.
Perceived student behavior | 20-weeks
  Assessed by teacher questionnaire on a 10-point scale from "No improvement" to "A great deal of improvement." Questions were averaged and higher scores indicated greater perceived student behavior.

CONTACTS AND LOCATIONS:
Overall Officials: John Cairney, PhD, Principal Investigator — University of Toronto and McMaster University
Locations (1):
- David Braley Health Sciences Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers

REFERENCES:
- [Background] Janssen I, Leblanc AG. Systematic review of the health benefits of physical activity and fitness in school-aged children and youth. Int J Behav Nutr Phys Act. 2010 May 11;7:40. doi: 10.1186/1479-5868-7-40. PMID 20459784
- [Background] Lubans D, Richards J, Hillman C, Faulkner G, Beauchamp M, Nilsson M, Kelly P, Smith J, Raine L, Biddle S. Physical Activity for Cognitive and Mental Health in Youth: A Systematic Review of Mechanisms. Pediatrics. 2016 Sep;138(3):e20161642. doi: 10.1542/peds.2016-1642. Epub 2016 Aug 19. PMID 27542849
- [Background] Ahn S, Fedewa AL. A meta-analysis of the relationship between children's physical activity and mental health. J Pediatr Psychol. 2011 May;36(4):385-97. doi: 10.1093/jpepsy/jsq107. Epub 2011 Jan 11. PMID 21227908
- [Background] Allison KR, Vu-Nguyen K, Ng B, Schoueri-Mychasiw N, Dwyer JJ, Manson H, Hobin E, Manske S, Robertson J. Evaluation of Daily Physical Activity (DPA) policy implementation in Ontario: surveys of elementary school administrators and teachers. BMC Public Health. 2016 Aug 8;16:746. doi: 10.1186/s12889-016-3423-0. PMID 27502505
- [Background] Pearlin LI, Lieberman MA, Menaghan EG, Mullan JT. The stress process. J Health Soc Behav. 1981 Dec;22(4):337-56. No abstract available. PMID 7320473
- [Background] Moilanen KL. The Adolescent Self-Regulatory Inventory: The development and validation of a questionnaire of short-term and long-term self-regulation. J Youth Adolesc. 2007;36:835-48.
- [Background] Goodman R, Meltzer H, Bailey V. The Strengths and Difficulties Questionnaire: a pilot study on the validity of the self-report version. Int Rev Psychiatry. 2003 Feb-May;15(1-2):173-7. doi: 10.1080/0954026021000046137. PMID 12745329
- [Background] Muris P, Meesters C, Eijkelenboom A, Vincken M. The self-report version of the Strengths and Difficulties Questionnaire: its psychometric properties in 8- to 13-year-old non-clinical children. Br J Clin Psychol. 2004 Nov;43(Pt 4):437-48. doi: 10.1348/0144665042388982. PMID 15530213
- [Background] Rosenberg M. Rosenberg Self-Esteem Scale. Accept Commit Ther. 1965.
- [Background] Duckworth AL, Quinn PD. Development and validation of the short grit scale (grit-s). J Pers Assess. 2009 Mar;91(2):166-74. doi: 10.1080/00223890802634290. PMID 19205937
- [Background] Lyubomirsky S, Lepper HS. A measure of subjective happiness: Preliminary reliability and construct validation. Soc Indic Res. 1999;46:137-155.
- [Background] Anderson-Butcher D, Conroy DE. Factorial and Criterion Validity of Scores of a Measure of Belonging in Youth Development Programs. Educ Psychol Meas. 2002;62:857-76.
- [Background] Crocker PR, Bailey DA, Faulkner RA, Kowalski KC, McGrath R. Measuring general levels of physical activity: preliminary evidence for the Physical Activity Questionnaire for Older Children. Med Sci Sports Exerc. 1997 Oct;29(10):1344-9. doi: 10.1097/00005768-199710000-00011. PMID 9346166
- [Background] Bandura A. Guide for constructing self-efficacy scales. Self-Effic Beliefs Adolesc. 2006;5.
- [Derived] Bremer E, Graham JD, Veldhuizen S, Cairney J. A program evaluation of an in-school daily physical activity initiative for children and youth. BMC Public Health. 2018 Aug 16;18(1):1023. doi: 10.1186/s12889-018-5943-2. PMID 30115054